CLINICAL TRIAL: NCT00929708
Title: A 4-week, Phase-II, Double-blind, Placebo-controlled, Randomised, Parallel-group, Multi-centre Study to Assess the Efficacy and Tolerability/Safety of Inhaled AZD3199 Once Daily Compared to 9 μg Formoterol Bid and Placebo in Patients With Moderate to Severe COPD
Brief Title: Efficacy of AZD3199 in Chronic Obstructive Pulmonary Disease (COPD) Patients
Acronym: GLAD
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: D0570C00003
Record Dates: First submitted 2009-06-26; First posted 2009-06-29 (Estimated); Results first posted 2014-01-17 (Estimated); Last update posted 2014-02-17 (Estimated); Status verified 2014-01

CONDITIONS: COPD
Keywords: COPD; Efficacy; Safety; Inhalation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Respiratory Aspiration | interventions — AZD-3199; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- 1 (Experimental): AZD3199 low dose
  Interventions: Drug: AZD3199
- 2 (Experimental): AZD3199 intermediate dose
  Interventions: Drug: AZD3199
- 3 (Experimental): AZD3199 high dose
  Interventions: Drug: AZD3199
- 4 (Active Comparator): Formoterol 2x4.5 microgram bid
  Interventions: Drug: formoterol
- 5 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: AZD3199 — Dry powder for inhalation, o.d., 4 weeks
  Arms: 1; 2; 3
Drug: formoterol — Dry powder for inhalation, b.i.d., 4 weeks
  Arms: 4
Drug: Placebo — Dry powder for inhalation, b.i.d., 4 weeks
  Arms: 5

SUMMARY:
The purpose of this study is to investigate the efficacy, safety and tolerability of 4 weeks treatment with AZD3199 in moderate to severe COPD.

ELIGIBILITY:
Inclusion Criteria:

* COPD
* Current or exsmokers, 10 pack years

Exclusion Criteria:

* Asthma
* Any clinically relevant abnormal findings at screening examinations
* Recent COPD exacerbation

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 329 (Actual)
Dates: Start 2009-06; Primary Completion 2010-03 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Piotr Kuna, Professor, Principal Investigator — University Hospital, Lodz, Poland
Locations (38):
- Bulgaria (5):
  - Research Site, Blagoevgrad
  - Research Site, Pleven
  - Research Site, Rousse
  - Research Site, Sofia
  - Research Site, Varna
- Canada (9):
  - Research Site, Moncton, New Brunswick
  - Research Site, St. John's, Newfoundland and Labrador
  - Research Site, Truro, Nova Scotia
  - Research Site, Greater Sudbury, Ontario
  - Research Site, Mississauga, Ontario
  - Research Site, Toronto, Ontario
  - Research Site, Pointe-Claire, Quebec
  - Research Site, Saint Romuald, Quebec
  - Research Site, Trois-Rivières, Quebec
- Japan (14):
  - Research Site, Yanagawa, Fukuoka
  - Research Site, Fukuyama, Hiroshima
  - Research Site, Chitose, Hokkaido
  - Research Site, Obihiro, Hokkaido
  - Research Site, Tomakomai, Hokkaido
  - Research Site, Hitachi, Ibaragi
  - Research Site, Naka-gun, Ibaraki
  - Research Site, Sendai, Miyagi
  - Research Site, Osaka, Osaka
  - Research Site, Toyonaka, Osaka
  - Research Site, Moriyama, Shiga
  - Research Site, Ōtsu, Shiga
  - Research Site, Machida, Tokyo
  - Research Site, Kitakyushu
- Poland (7):
  - Research Site, Bialystok
  - Research Site, Gorzow Wlkp
  - Research Site, Lodz
  - Research Site, Lublin
  - Research Site, Poznan
  - Research Site, Szczecin
  - Research Site, Tarnów
- Russia (3):
  - Research Site, Moscow
  - Research Site, Novosibirsk
  - Research Site, Saint Petersburg

REFERENCES:
- [Derived] Kuna P, Ivanov Y, Trofimov VI, Saito T, Beckman O, Bengtsson T, Jorup C, Maltais F. Efficacy and safety of AZD3199 vs formoterol in COPD: a randomized, double-blind study. Respir Res. 2013 Jun 3;14(1):64. doi: 10.1186/1465-9921-14-64. PMID 23731768

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study has been performed at 53 centres in Bulgaria, Canada, Japan, Poland and Russian Federation. The recruitment period was between 16 June 2009 and 8 January 2010.
Groups:
- AZD3199 200 Mcg od: 2 x AZD3199 Turbuhaler 100 mcg (morning) + 2 x placebo Turbuhaler (evening)
- AZD3199 400 Mcg od: 2 x AZD3199 Turbuhaler 200 mcg (morning) + 2 x placebo Turbuhaler (evening)
- AZD3199 800 Mcg od: 2 x AZD3199 Turbuhaler 400 mcg (morning) + 2 x placebo Turbuhaler (evening)
- Formoterol 9 Mcg Bid: 2 x Oxis Turbuhaler 4.5 mcg (morning) + 2 x Oxis Turbuhaler 4.5 mcg (evening)
- Placebo: 2 x placebo Turbuhaler (morning) + 2 x placebo Turbuhaler (evening)
Period: Overall Study
Arm/Group | AZD3199 200 Mcg od | AZD3199 400 Mcg od | AZD3199 800 Mcg od | Formoterol 9 Mcg Bid | Placebo
Started | 65 | 69 | 65 | 67 | 63
Completed | 61 | 66 | 62 | 61 | 57
Not Completed | 4 | 3 | 3 | 6 | 6
Not completed — Protocol Violation | 2 | 1 | 1 | 1 | 1
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 2 | 1
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 3
Not completed — Physician Decision | 0 | 2 | 2 | 2 | 1
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | AZD3199 200 Mcg od | AZD3199 400 Mcg od | AZD3199 800 Mcg od | Formoterol 9 Mcg Bid | Placebo | Total
Number analyzed (Participants) | 65 | 69 | 65 | 67 | 63 | 329
Age, Continuous [Mean (Full Range); unit: Years] | 62.4 [45 to 81] | 63.8 [40 to 82] | 65.3 [41 to 92] | 64.1 [47 to 77] | 64.8 [46 to 84] | 63.85 [62.4 to 65.3]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18 | 16 | 20 | 16 | 12 | 82
  Male | 47 | 53 | 45 | 51 | 51 | 247

OUTCOME MEASURES:

1. Primary Outcome: FEV1, E0-4; the Average Value at Visit 5 From Before to 4 Hours After Morning Dose (Peak Effect)
Description: change from baseline
Time Frame: 0,5 min, 15 min, 60 min, 2 h, 4 h
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | AZD3199 200 Mcg od | AZD3199 400 Mcg od | AZD3199 800 Mcg od | Formoterol 9 Mcg Bid | Placebo
Number analyzed (Participants) | 61 | 66 | 63 | 62 | 57
Litre | 0.21 (0.33) | 0.17 (0.31) | 0.14 (0.27) | 0.16 (0.22) | 0.03 (0.25)

2. Primary Outcome: FEV1, E24-26; the Average Value at Visit 5 Between 24 and 26 Hours Following the Morning Dose (Trough Effect)
Description: change from baseline
Time Frame: 24h, 26h
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | AZD3199 200 Mcg od | AZD3199 400 Mcg od | AZD3199 800 Mcg od | Formoterol 9 Mcg Bid | Placebo
Number analyzed (Participants) | 61 | 66 | 62 | 62 | 57
Litre | 0.11 (0.31) | 0.12 (0.28) | 0.11 (0.25) | 0.03 (0.23) | 0.01 (0.24)

3. Secondary Outcome: Cmax; the Highest Plasma Concentration of AZD3199 Measured
Description: PK is only measured for AZD3199
Time Frame: 0,15 min, 1, 4 and 24 hours post dose
Population: AZD3199 plasma data were available for 178 of the 199 randomized patients, but data from 2 patients in AZD3199 200 mcg group were excluded from analysis because most of the values were below LOQ.
Measure: Geometric Mean (Full Range); unit: nmol/L
Arm/Group | AZD3199 200 Mcg od | AZD3199 400 Mcg od | AZD3199 800 Mcg od | Formoterol 9 Mcg Bid | Placebo
Number analyzed (Participants) | 53 | 64 | 59 | 0 | 0
nmol/L | 1.14 [0.03 to 3.6] | 1.88 [0.05 to 9.8] | 4.01 [0.12 to 18.2] |  |

4. Secondary Outcome: AUC0-24; Area Under the Plasma Concentration Curve From Zero to 24 Hours After Dose
Description: PK is only measured for AZD3199
Time Frame: 0,15 min, 1, 4 and 24 hours post dose
Population: as for outcome 3
Measure: Geometric Mean (Full Range); unit: nmol*h/L
Arm/Group | AZD3199 200 Mcg od | AZD3199 400 Mcg od | AZD3199 800 Mcg od | Formoterol 9 Mcg Bid | Placebo
Number analyzed (Participants) | 53 | 64 | 59 | 0 | 0
nmol*h/L | 4.83 [0.4 to 20.8] | 8.69 [0.7 to 54.1] | 14.82 [1.4 to 76.3] |  |

5. Secondary Outcome: FEV1 Post Salbutamol Inhalation
Description: Mean value of FEV1 pre and post salbutamol at visit 2 and visit 5
Time Frame: Baseline (visit 2) and 26 h after the last morning dose (visit 5).
Measure: Mean (Standard Deviation); unit: Litre
Arm/Group | AZD3199 200 Mcg od | AZD3199 400 Mcg od | AZD3199 800 Mcg od | Formoterol 9 Mcg Bid | Placebo
Number analyzed (Participants) | 61 | 62 | 61 | 61 | 54
Litre | 0.060 (0.306) | 0.073 (0.358) | 0.077 (0.238) | 0.048 (0.260) | 0.018 (0.215)

6. Secondary Outcome: Total Number of Reliever Medication Inhalations Per 24h
Description: Change from run-in
Time Frame: During day (from rising from bed until going to bed) and night (from going to bed until rising from bed) at visit 1 to visit 5 (24h), up to 4 weeks.
Measure: Mean (Standard Deviation); unit: Number of reliver inh.
Arm/Group | AZD3199 200 Mcg od | AZD3199 400 Mcg od | AZD3199 800 Mcg od | Formoterol 9 Mcg Bid | Placebo
Number analyzed (Participants) | 64 | 66 | 64 | 63 | 60
Number of reliver inh. | -0.96 (1.85) | -1.23 (1.96) | -1.15 (1.55) | -0.66 (1.40) | -0.23 (1.58)

7. Secondary Outcome: Total AstraZeneca COPD Symptoms Scores (Included Breathlessness, Chest Tightness, Cough and Night-time Awakenings)
Description: Score on a scale 5-point Likert-type scale, ranging from 0 (none) to 4 (severe) for each symptom, total score is the sum of each symptom ranged from 0 to 16. Change from run-in.
Time Frame: Daily, during run-in and treatment
Measure: Mean (Standard Deviation); unit: total score
Arm/Group | AZD3199 200 Mcg od | AZD3199 400 Mcg od | AZD3199 800 Mcg od | Formoterol 9 Mcg Bid | Placebo
Number analyzed (Participants) | 64 | 66 | 64 | 63 | 60
total score | -0.96 (1.34) | -0.91 (1.65) | -1.21 (1.53) | -0.56 (1.83) | -0.43 (1.61)

8. Secondary Outcome: Overall Mean CCQ (Clinical COPD Questionnaire)
Description: Change from baseline to treatment in score. The total scores vary between 0 (never/not limited at all) to 6 (almost all the time/totally limited). The data below represent the average of week 1,2,4 minus week 0.
Time Frame: Mean over week 0, mean over week 1, mean over week 2, and mean over week 4
Measure: Mean (Standard Deviation); unit: score on scale
Arm/Group | AZD3199 200 Mcg od | AZD3199 400 Mcg od | AZD3199 800 Mcg od | Formoterol 9 Mcg Bid | Placebo
Number analyzed (Participants) | 64 | 69 | 64 | 66 | 61
score on scale | -0.39 (0.49) | -0.29 (0.65) | -0.39 (0.54) | -0.35 (0.65) | -0.10 (0.70)

9. Secondary Outcome: Total Score SGRQ-C (St George's Respiratory Questionnaire for COPD)
Description: The total score is calculated using all questions including their weights and scores range from 0 (perfect health) to 100 (worst possible state)
Time Frame: At baseline (visit 2) and after 4 weeks of treatment (visit 5).
Measure: Mean (Standard Deviation); unit: Score
Arm/Group | AZD3199 200 Mcg od | AZD3199 400 Mcg od | AZD3199 800 Mcg od | Formoterol 9 Mcg Bid | Placebo
Number analyzed (Participants) | 59 | 66 | 61 | 58 | 53
Score | -5.10 (13.67) | -8.17 (12.18) | -5.01 (10.69) | -5.16 (10.88) | -2.35 (12.98)

ADVERSE EVENTS:
Arm/Group | AZD3199 200 Mcg od | AZD3199 400 Mcg od | AZD3199 800 Mcg od | Formoterol 9 Mcg Bid | Placebo
Serious Adverse Events (participants affected / at risk) | 1/65 | 4/69 | 0/65 | 3/67 | 2/63
Other Adverse Events (participants affected / at risk) | 1/65 | 8/69 | 7/65 | 4/67 | 3/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | AZD3199 200 Mcg od (N=65) | AZD3199 400 Mcg od (N=69) | AZD3199 800 Mcg od (N=65) | Formoterol 9 Mcg Bid (N=67) | Placebo (N=63)
Chroniv obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Colitis ishaemic (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Hypertensive crisis (Vascular disorders) | 0 | 0 | 0 | 0 | 1
Macular degeneration (Eye disorders) | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0 | 0
Circulatory collapse (Vascular disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | AZD3199 200 Mcg od (N=65) | AZD3199 400 Mcg od (N=69) | AZD3199 800 Mcg od (N=65) | Formoterol 9 Mcg Bid (N=67) | Placebo (N=63)
Nasopharyngitis (Infections and infestations) | 1 | 4 | 3 | 2 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 4 | 2 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
An Investigator agrees to provide a copy of the publication to AZ for review at least 60 days in advance of submission for publication. Investigators in multicenter (MC) studies agree to postpone MC publications until the earlier of the date of the first AZ-authorized MC publication or a period up to 18 months from study completion at all sites. AZ has the right to request delays: up to 60 days for confidential information, and an additional 90 days to protect intellectual property.